CLINICAL TRIAL: NCT04326348
Title: A Single-arm, Open-label, Phase I Study of TQ05105 Tablets in Subjects With Hemophagocytic Lymphohistiocytosis.
Brief Title: A Study of TQ05105 Tablets in Subjects With Hemophagocytic Lymphohistiocytosis（HLH）
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-I-02
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-03

CONDITIONS: Hemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ05105 Tablet (Experimental): TQ05105 tablet administered orally once. Then TQ05105 tablet administered orally, twice daily in 28-day cycle after 3 days of first administration.
  Interventions: Drug: TQ05105

INTERVENTIONS:
Drug: TQ05105 — TQ05105 is a JAK2 inhibitor.

SUMMARY:
This is a phase I study of TQ05105 tablets in subjects with Hemophagocytic Lymphohistiocytosis.TQ05105 is a JAK2 inhibitors and can be used to treat JAK2 target-related diseases. The activation of the JAK/STAT pathway is related to abnormal proliferation, obstruction of apoptosis, and differentiation disorder of leukemia cells which is caused by genetic abnormalities and viral infection.

ELIGIBILITY:
Inclusion Criteria:

* 1.18 years and older; Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3; Life expectancy ≥ 3 months.

  2. Diagnosed as new or relapsed HLH according to the HLH-2004 criteria. 3.Has received other treatments for HLH before two weeks ago, surgery before four weeks ago.

  4. Adequate laboratory indicators. 5. No pregnant or breastfeeding women, and a negative pregnancy test. 6. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization. With exception of non-melanoma, skin cancer, and carcinoma in situ.

  2. Has participated in other anticancer drug clinical trials within 4 weeks. 3. Has multiple factors affecting oral medication. 4. Has drug abuse history that unable to abstain from or mental disorders. 5. Has active hepatitis B or C, or immunodeficiency. 6. Diagnosed as hepatic failure. 7. Has arteriovenous thrombosis events within 4 weeks. 8. Has active bleeding, or a persistent decrease in hemoglobin. 9. Has received long-term and large-dose glucocorticoids or other immunosuppressive drugs within 28 days before signed the informed consent form.

  10. Has uncontrolled cardiovascular disease. 11. Has uncontrolled hypertension. 12. Has serious systemic infections. 13. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Baseline up to 28 days
  DLT defined as any of the events occurring during the study related to drugs.
Maximal tolerance dose (MTD) | Baseline up to 28 days
  MTD defined as the highest dose level at which less than or equal to 2 of 6 subjects experience dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Cmax | Hour 0, 5, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 11, 24 hours post-dose on single dose; Hour 0 of day 1,day 3,day5, day 6 on multiple dose and hour0, 5, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 11 hours post-dose on multiple dose of day 28.
  Cmax is the maximum plasma concentration of TQ05105 or metabolite(s).
Tmax | Hour 0, 5, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 11, 24 hours post-dose on single dose; Hour 0 of day 1,day 3,day5, day 6 on multiple dose and hour0, 5, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 11 hours post-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQ05105 by assessment of time to reach maximum plasma concentration.
AUC0-t | Hour 0, 5, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 11, 24 hours post-dose on single dose; Hour 0 of day 1,day 3,day5, day 6 on multiple dose and hour0, 5, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 11 hours post-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQ05105 by assessment of area under the plasma concentration time curve from zero to infinity.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China